CLINICAL TRIAL: NCT02785692
Title: Preoperative IMRT for Soft Tissue Sarcoma of the Extremities and Trunk: Low Rate of Wound Complications
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator has left the Institution
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-00100
Record Dates: First submitted 2016-05-16; First posted 2016-05-30 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Sarcoma
Keywords: soft tissue sarcoma; IMRT and sarcoma; preoperative highly conformal radiation therapy; soft tissue sarcoma and wound healing; postoperative complications; treatment tolerance of soft tissue IMRT
MeSH Terms: conditions — Sarcoma; Postoperative Complications | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Combined Radiation/ Surgery: All patients treated with combined radiotherapy and surgery at Balgrist University Hospital and University Hospital Zurich
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — preoperative Radiotherapy/ IMRT

SUMMARY:
Postoperative wound healing complications following preoperative radiotherapy represent a severe problem in the treatment of malignant soft tissue tumors, and are reported to be 34% and more. The literature discusses intensely the advantages and disadvantages of this multimodal treatment concept and there are different opinions. The Canadian prospective randomized NCIC SR2 trial showed increased wound complication rates in the study arm receiving preoperative radiation. The Sarcoma Center Zurich pursues mainly this treatment concept and the results shall now be analysed and published. The approach is to show that not only the complication rates are comparable to international bench marks, but also the (still intermediate time) local control rates.

DETAILED DESCRIPTION:
Introduction: The Canadian prospective randomized NCIC SR2 trial tested the sequence of radiation and surgery for soft tissue sarcoma of the extremities. Similar disease control rates following pre- versus postoperative non-intensity modulated radiation therapy (non-IMRT) was found, with increased wound complications (17% vs 35%) in the preoperative radiation arm, [95% CI 5-30], p=0·01).

The investigators assessed a single center preoperative IMRT (or IMRT-equivalent highly conformal three dimensional conventional RT (3DcRT)) cohort with respect to the wound complication rate (WCR). The hypothesis was that a lower WCR rate was achieved in the era of IMRT as compared to the non-IMRT era when the Canadian Trial was conducted.

Methods: 67 consecutive patients irradiated with 50Gy in 25 fractions between 3/2008-3/2016 with preoperative IMRT (n=48, 72%) or highly conformal IMRT-equivalent 3DcRT dose distribution (n=19, 28%) were assessed. All patients were previously discussed at the weekly interdisciplinary sarcoma board of the Sarcoma Center Zurich.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a malignant soft tissue tumour
* Patients who underwent preoperative radiotherapy at the department of radiation oncology, University Hospital Zurich (USZ)
* Surgical treatment at Balgrist University Hospital between 2007 and 2016

Exclusion Criteria:

* Vulnerability
* Previous chemotherapy
* Previous radiotherapy on the affected site
* Patient's wish

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 67 patients with histological proven malignant soft tissue sarcomas who underwent preoperative radiotherapy followed by surgical tumor resection
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Major and minor wound healing complications | through study completion, minimum 6 weeks post surgery

SECONDARY OUTCOMES:
Local and metastatic disease control based on imaging such as CT scans and MRI | maximum 10 years post surgery
Overall survival at the latest point of follow- up | maximum 10 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Fuchs, Prof. MD PhD, Study Chair — Balgrist University Hospital
Locations (2):
- Switzerland (2):
  - Balgrist University Hospital, Zurich
  - University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: No